CLINICAL TRIAL: NCT06529081
Title: Assessment of Radiotherapy Strategies for Use in Combined Treatment of Small-cell Lung Cancer at the Stage of Extensive Disease - a Research Experiment
Brief Title: Radiotherapy Strategies for Use in Combined Treatment of Small-cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copernicus Memorial Hospital (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Łukasz Kuncman, Principal Investigator, Copernicus Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/ABM/01/00040
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Small Cell Lung Carcinoma; Extensive Disease; Chemo-immunotherapy; Radiotherapy; Durvalumab; Atezolizumab; Immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Treatment (No Intervention): PDL1/PD1 immunotherapy (durvalumab or atezolozumab - according to the SmPC) after chemo-immunotherapy based on platinum compounds.
- Standard Treatment with Palliative Radiotherapy (Experimental)
  Interventions: Radiation: Palliative Radiotherapy
- Standard Treatment with Radical/Ablative Radiotherapy (Experimental)
  Interventions: Radiation: Radical/Ablative Radiotherapy

INTERVENTIONS:
Radiation: Palliative Radiotherapy — Standard treatment with added consolidative radiotherapy to the chest area and possibly metastatic lesions (if indicated) in doses and for palliative indications (total dose of 30 Gy in 10 daily doses of 3 Gy each).
  Arms: Standard Treatment with Palliative Radiotherapy
Radiation: Radical/Ablative Radiotherapy — Standard treatment with added radical/ablative radiotherapy (total dose of 45 Gy in 15 daily fractions of 3 Gy to the chest area and total dose of 24 Gy administered in single fractions of 8 Gy every 2-3 days to the metastatic lesions) to the chest area and all metastatic lesions.
  Arms: Standard Treatment with Radical/Ablative Radiotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of radiotherapy as part of the combined treatment approach for patients diagnosed with histopathologically confirmed small cell lung cancer (SCLC) in the advanced stage of extensive disease (ED) who are undergoing chemo-immunotherapy. The planned study aims to assess the impact of incorporating consolidative radiotherapy into the treatment strategy, focusing on residual changes following chemo-immunotherapy (during immunotherapy) and its effect on progression-free survival.

This research experiment will be conducted as a randomized multi-center study, comprising the following treatment arms:

* Arm I: Continuation of standard of care - PDL1/PD1 immunotherapy (durvalumab or atezolozumab) after chemo-immunotherapy based on platinum compounds;
* Arm II: Standard of care, followed by consolidating radiotherapy of the chest area and possibly metastases (if indicated) in doses and for palliative indications (total dose of 30 Gy in 10 daily doses of 3 Gy each);
* Arm III: Standard of care, followed by consolidating radiotherapy in the radical/ablative doses (total dose of 45 Gy delivered in 15 daily fractions of 3 Gy for the chest area, and total dose of 24 Gy in single fractions of 8 Gy administered every 2-3 days for the metastatic lesions) of the chest area and all metastatic lesions.

Additionally, as part of routine weekly blood collections, an extra volume of 10 ml of blood will be collected. This additional blood sample will be obtained before starting radiotherapy, during each week of radiotherapy (maximum three collections), and at the time of disease progression (one collection), resulting in a total of five extra samples. The collected blood will be prepared, stored and used for circulating tumor DNA (ctDNA) testing, according to the protocol. The ctDNA analysis data will be utilized as a potential marker to determine the time to progression and assess the benefits derived from the administered radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological confirmation of small cell lung cancer based on histological or cytological examination.
* Primary clinical stage: Extensive stage of the disease according to VASLG classification or stage IV according to TNM classification.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 prior to randomization.
* Partial response (PR) or stable disease (SD) to platinum-based doublet chemotherapy with durvalumab or atezolizumab based on restaging (positron emission tomography [PET]/computed tomography [CT] or CT or magnetic resonance imaging [MRI]).
* Ability to undergo radiotherapy at a total dose of 45 Gy in 15 daily fractions of 3 Gy to the chest area and a total dose of 24 Gy administered in single fractions every 2-3 days of 8 Gy to the metastatic lesions.
* Clinical control of brain metastases (prior whole-brain irradiation at any stage is acceptable before study entry).
* Measurable residual disease after chemioimmunotherapy (according to RECIST 1.1 solid tumor response assessment criteria) or in case of CR/PR presence of tumor lesions not classified as measurable.
* Volume and number (up to 10) of metastatic lesions allowing for radiotherapy in doses according to the study protocol.
* Absence of clinically significant and uncontrolled co-morbidities with pharmacological treatment.
* Absence of active autoimmune diseases except for diabetes, hypothyroidism, psoriasis, eczema, lichen planus, and vitiligo.
* Adequate hematopoietic function allowing treatment with atezolizumab or durvalumab, according to the current SmPC (Summary of Product Characteristics).
* Renal and hepatic function allowing treatment according to the current SmPC for atezolizumab or durvalumab.

Exclusion Criteria:

* Age under 18 years old.
* Premenopausal women who do not accept the need for effective contraception during radiotherapy and/or chemotherapy/immunotherapy.
* Individuals excluded from participation in a medical experiment based on Article 23A(1) of the Act on the Profession of Physician and Pharmacist.
* Coexistence of other uncontrolled malignant neoplasms.
* Contraindications to the use of atezolizumab or durvalumab as specified in the SmPC.
* Grade 2 or greater CTCAE v.5 pneumonitis secondary to immunotherapy.
* Participation in another clinical trial during the study.
* Prior chest radiotherapy that precludes safe administration of radiotherapy according to the study protocol. Prior palliative radiotherapy to metastatic sites is acceptable before study entry if clinically indicated as determined by the physician.
* Contraindications to radiotherapy according to the approved protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to RECIST 1.1 imaging criteria or patient death. | 12 months after last patient entry
  The assessment of the impact of consolidative (radical/palliative) radiotherapy on residual post-chemoimmunotherapy (during immunotherapy) lesions on progression-free survival (PFS).

SECONDARY OUTCOMES:
Overall survival. | At the end of the study (an average of 1 year after last patient entry).
Treatment toxicity (incidence of Grade 3 toxicity according to CTCAE v.5). | At the end of the study (an average of 1 year after last patient entry).
Site of progression (primary lesions [present at baseline]/new lesions). | At the end of the study (an average of 1 year after last patient entry).
Objective response rate (ORR). | At the end of the study (an average of 1 year after last patient entry).
Response rate in nonirradiated lesions. | At the end of the study (an average of 1 year after last patient entry).

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Kuncman, PhD, Principal Investigator — Department of Radiotherapy, Copernicus Memoriał Hospital in Łódź, Poland
Locations (2):
- Poland (2):
  - Center of Oncology of the Lublin Region St. Jana z Dukli in Lublin, Lublin
  - Copernicus Memorial Hospital in Łódź, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faivre-Finn C, Snee M, Ashcroft L, Appel W, Barlesi F, Bhatnagar A, Bezjak A, Cardenal F, Fournel P, Harden S, Le Pechoux C, McMenemin R, Mohammed N, O'Brien M, Pantarotto J, Surmont V, Van Meerbeeck JP, Woll PJ, Lorigan P, Blackhall F; CONVERT Study Team. Concurrent once-daily versus twice-daily chemoradiotherapy in patients with limited-stage small-cell lung cancer (CONVERT): an open-label, phase 3, randomised, superiority trial. Lancet Oncol. 2017 Aug;18(8):1116-1125. doi: 10.1016/S1470-2045(17)30318-2. Epub 2017 Jun 20. PMID 28642008
- [Background] Horn L, Mansfield AS, Szczesna A, Havel L, Krzakowski M, Hochmair MJ, Huemer F, Losonczy G, Johnson ML, Nishio M, Reck M, Mok T, Lam S, Shames DS, Liu J, Ding B, Lopez-Chavez A, Kabbinavar F, Lin W, Sandler A, Liu SV; IMpower133 Study Group. First-Line Atezolizumab plus Chemotherapy in Extensive-Stage Small-Cell Lung Cancer. N Engl J Med. 2018 Dec 6;379(23):2220-2229. doi: 10.1056/NEJMoa1809064. Epub 2018 Sep 25. PMID 30280641
- [Background] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Use of thoracic radiotherapy for extensive stage small-cell lung cancer: a phase 3 randomised controlled trial. Lancet. 2015 Jan 3;385(9962):36-42. doi: 10.1016/S0140-6736(14)61085-0. Epub 2014 Sep 14. PMID 25230595
- [Background] Goldman JW, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Garassino MC, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Thiyagarajah P, Jiang H, Paz-Ares L; CASPIAN investigators. Durvalumab, with or without tremelimumab, plus platinum-etoposide versus platinum-etoposide alone in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): updated results from a randomised, controlled, open-label, phase 3 trial. Lancet Oncol. 2021 Jan;22(1):51-65. doi: 10.1016/S1470-2045(20)30539-8. Epub 2020 Dec 4. PMID 33285097
- [Background] Gore EM, Hu C, Sun AY, Grimm DF, Ramalingam SS, Dunlap NE, Higgins KA, Werner-Wasik M, Allen AM, Iyengar P, Videtic GMM, Hales RK, McGarry RC, Urbanic JJ, Pu AT, Johnstone CA, Stieber VW, Paulus R, Bradley JD. Randomized Phase II Study Comparing Prophylactic Cranial Irradiation Alone to Prophylactic Cranial Irradiation and Consolidative Extracranial Irradiation for Extensive-Disease Small Cell Lung Cancer (ED SCLC): NRG Oncology RTOG 0937. J Thorac Oncol. 2017 Oct;12(10):1561-1570. doi: 10.1016/j.jtho.2017.06.015. Epub 2017 Jun 23. PMID 28648948
- [Background] Timmerman R. A Story of Hypofractionation and the Table on the Wall. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):4-21. doi: 10.1016/j.ijrobp.2021.09.027. No abstract available. PMID 34919882
- [Background] Herbreteau G, Langlais A, Greillier L, Audigier-Valette C, Uwer L, Hureaux J, Moro-Sibilot D, Guisier F, Carmier D, Madelaine J, Otto J, Souquet PJ, Gounant V, Merle P, Molinier O, Renault A, Rabeau A, Morin F, Denis MG, Pujol JL. Circulating Tumor DNA as a Prognostic Determinant in Small Cell Lung Cancer Patients Receiving Atezolizumab. J Clin Med. 2020 Nov 27;9(12):3861. doi: 10.3390/jcm9123861. PMID 33261056
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Derived] Kuncman L, Fijuth J, Tworek D, Sierko E, Cisek P, Maslowski M, Lisik-Habib M, Orzechowska M, Galwas-Kliber K, Antczak A, Chmielewska I, Ziolkowska B, Kurczewska-Michalak M, Kuznicki W, Jedrzejczak N, Ranoszek K, Bilski M. Radiotherapy(R) Integration(I) Strategy for Small(S)-Cell Lung Cancer in Extensive(E) Stage (RISE) with up to 10 metastases- a study protocol of a randomized phase II trial. BMC Cancer. 2025 Jan 24;25(1):142. doi: 10.1186/s12885-025-13552-y. PMID 39856583

DOCUMENTS (1):
  • Informed Consent Form (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT06529081/ICF_000.pdf